CLINICAL TRIAL: NCT04651049
Title: Influence of Systemic Propranolol Treatment on the Physical Development of Paediatric Patients With Infantile Hemangiomas
Brief Title: Systemic Propranolol for the Treatment of Paediatric Patients With Infantile Hemangiomas
Status: Completed | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: LiuSH
Record Dates: First submitted 2020-11-18; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-08

CONDITIONS: Infantile Haemangiomas
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Propranolol treatment group
  Interventions: Drug: propranolol

INTERVENTIONS:
Drug: propranolol — This retrospective study included 128 patients treated with oral propranolol at a dose of 2.0 mg/kg per day.
Device:

SUMMARY:
This is retrospective study. The patients treated with oral propranolol at a dose of 2.0 mg/kg per day. Growth parameters (height and weight) were measured at the beginning, the end of treatment and 2 years after treatment. The weight-for-age Z-score (WAZ), height-for-age Z-score (HAZ) and weight-for-height Z-score (WHZ) calculated by the WHO Anthro software were used to assess physical development, and the WHO Child Growth Standards were used as the standards.

ELIGIBILITY:
Inclusion Criteria:

* IHs diagnosed by medical history and physical examination
* no previous treatment with other medications

Exclusion Criteria:

* a history or risk of asthma, reactive airway disease, impaired renal or liver function, heart defects or arrhythmia, hypotension and hypersensitivity to propranolol
* Infants who did not adhere to the treatments or attend follow-up visits
* Infants with other known risk factors for developmental delay or growth restriction, such as prematurity, small for gestational age, or other major congenital malformations, were also excluded
* No other treatment was used during the oral propranolol course

Ages: 2 Weeks to 54 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Overall, 52 males and 76 females, with a male-to-female ratio of 1:1.46, were included in this study. Of the 128 patients, 16 (12.5%) were born prematurely. The median age at the start of propranolol therapy was 3.75 months (0.5-12.5 months). Propranolol was administered for a median duration of 10.52 months (2-24 months).
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change on the height of the patients | at the beginning of the treatment, at the end of treatment and 2 years after the treatment
  we recorded the height of the patients in meters.
Change on the weight of the patients | at the beginning of the treatment, at the end of treatment and 2 years after the treatment
  we recorded the weight of the patients in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Shaohua Liu, Dr., Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen ZY, Wang QN, Zhu YH, Zhou LY, Xu T, He ZY, Yang Y. Progress in the treatment of infantile hemangioma. Ann Transl Med. 2019 Nov;7(22):692. doi: 10.21037/atm.2019.10.47. PMID 31930093
- [Result] Hoeger PH, Harper JI, Baselga E, Bonnet D, Boon LM, Ciofi Degli Atti M, El Hachem M, Oranje AP, Rubin AT, Weibel L, Leaute-Labreze C. Treatment of infantile haemangiomas: recommendations of a European expert group. Eur J Pediatr. 2015 Jul;174(7):855-65. doi: 10.1007/s00431-015-2570-0. Epub 2015 May 29. PMID 26021855